CLINICAL TRIAL: NCT01177787
Title: Clinical Efficacy of Local Fat Reduction on the Thigh of Korean Women Through Cryolipolysis
Brief Title: Clinical Efficacy of Cryolipolysis on the Fat of Thigh in Korean Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonik Trade Company, Korea (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Wonik201007
Record Dates: First submitted 2010-07-28; First posted 2010-08-09 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-04

CONDITIONS: Lipolysis; Cryotherapy Effect
Keywords: cryolipolysis; fat; thigh; Korean women
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- zeltiq (Active Comparator): Cryolipolysis had been done for 1 hour on ipsilateral thigh fat through Zeltiq machine.
  Interventions: Device: zeltiq
- electrical stimulation (Sham Comparator): Lipolysis had been done for 30 minutes on controlateral thigh fat through amplitude modulated frequency.
  Interventions: Device: electrical stimulation

INTERVENTIONS:
Device: zeltiq — Cryolipolysis had been conducted for targeted fat area on thigh for 1 hour through Zeltiq machine made in Zeltiq Aesthetics.
  Other Names: zeltiq, cryolipolysis
  Arms: zeltiq
Device: electrical stimulation — Lipolysis would be done on controlateral thigh for 30 minutes through 3000 Hz- amplitude modulated frequency.
  Other Names: electrical frequency
  Arms: electrical stimulation

SUMMARY:
The aim of this study is to evaluate the clinical efficacy of reduction of local fat on ipsilateral thigh through cryolipolysis (zeltiq) and controlateral thigh using by amplitude modulated frequency (conventional) method.

DETAILED DESCRIPTION:
Cryolipolysis is a new concept to reduce fat since Zeltiq machine had been introduced several years ago. Several different trials such as high frequency, liposuction and chemical lipolysis to remove fat had been emerged and tried. Therefore, we would like to know the clinical efficacy of cryolipolysis through comparative experiment with former frequency method on each thigh on healthy Korean women.

Healthy premenopausal women who want to reduce the fat on thigh were included. 28 healthy volunteered women recruited for this study, 15 subjects among participated after interviewing, sampling their metabolic variables at initial visit. A total of 15 subjects would be investigated through food diary(24hour), femoral CT, anthropometric, metabolic variables at initial, 4th, 12th week. Histological examination under skin(initial and 12th week), questionnaire(4th, 12th week) for satisfaction, adverse events would be monitored during 3 month.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal healthy women
* subjects with body mass index >= 18.
* subjects with visible fat on both thigh
* subjects to understand and agree to this study protocol

Exclusion Criteria:

* subjects with cryoglobulinemia, cold urticaria, or paroxysmal cold hemogobulinemia
* subjects with pregnancy or lactation within 6 months or next 3 months
* subjects with any laboratory, or metabolic abnormalities
* uncooperative subjects to comply with the study protocol
* women taking any medication over 6 months
* subjects with menstrual irregularities
* subjects to change over 10% of the former weight within the past 6 months - any procedure such as liposuction, or another surgical procedure or mesotherapy to reduce fat within 6 months
* subjects with any dermatologic abnormalities on the target area (thigh)
* subjects with any injection into the area of intended treatment (e.g. cortisone) within 6 months

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2010-09-30 (Actual); Study Completion 2010-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Rae Lee, MD.PhD., Principal Investigator — Director of Bariatric medicine, Family Medicine, Hong-Ik General Hospital
Locations (1):
- Bariatric clinic/Family medicine, Hong-Ik General Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KR Lee. Clinical Efficacy of Fat Reduction on the Thigh of Korean Women through CryolipolysisJ Obes Weight Loss Ther 2013, 3:6
- See also: obesity & weight loss therapy web site — http://dx.doi.org/10.4172/2165-7904.1000203
- Available data/document: Individual Participant Data Set — http://dx.doi.org/10.4172/2165-7904.1000203

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two arm, but same group. Electrical Stimulation on Rt thigh versus Zeltiq Application on Left thigh.
Groups:
- Zeltiq on Left/ Electrical Stimulation on Right Thigh: Cryolipolysis had been done for 1 hour on ipsilateral thigh fat through Zeltiq machine.
  zeltiq: Cryolipolysis had been conducted for targeted fat area on thigh for 1 hour through Zeltiq machine made in Zeltiq Aesthetics.
  Lipolysis had been done for 30 minutes on controlateral thigh fat through amplitude modulated frequency.
  electrical stimulation: Lipolysis would be done on controlateral thigh for 30 minutes through 3000 Hz- amplitude modulated frequency.
Period: Clinical Efficacy of Cryolipolysis
Arm/Group | Zeltiq on Left/ Electrical Stimulation on Right Thigh
Started | 28
Completed | 28
Not Completed | 0
Period: Cryolipolysis on Thigh
Arm/Group | Zeltiq on Left/ Electrical Stimulation on Right Thigh
Started | 28
Completed | 14
Not Completed | 14
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 9
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: A total of 14 subjects were completed this study.
Groups:
- Zeltiq on Left/Electrical Stimulation on Rt: Cryolipolysis had been done for 1 hour on ipsilateral thigh fat through Zeltiq machine.
  zeltiq: Cryolipolysis had been conducted for targeted fat area on thigh for 1 hour through Zeltiq machine made in Zeltiq Aesthetics.
  Lipolysis had been done for 30 minutes on controlateral thigh fat through amplitude modulated frequency.
  electrical stimulation: Lipolysis would be done on controlateral thigh for 30 minutes through 3000 Hz- amplitude modulated frequency.
Arm/Group | Zeltiq on Left/Electrical Stimulation on Rt
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.57 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Cross Sectional Area of Fat in Both Thighs
Description: reduction of fat amounts on both thighs measured by computerizing tomography
Time Frame: 4 weeks
Population: Cross sectional areas of both thighs at initial visit
Measure: Mean (Standard Deviation); unit: millimeters squares
Groups:
- Cross Sectional Area on Left Thigh: Cross Sectional Area (mm squares) on Left Thigh by CT
- Cross Sectional Area on Right Thigh: Cross Sectional Area (mm squares) on Rt thigh by CT
Arm/Group | Cross Sectional Area on Left Thigh | Cross Sectional Area on Right Thigh
Number analyzed (Participants) | 14 | 14
millimeters squares | -420.25 (3099.55) | -28.53 (3526.21)

2. Primary Outcome: Change of the Girths in Both Thighs
Description: Mean differences of the circumferences of both thighs measured by inches
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: inches
Groups:
- Zeltiq on Left: Cryolipolysis using by Zeltiq for 1 hour
- Electrical Stimulation on Right Side Thigh: The radio frequency method was applied on right thigh (control side) as sham procedure for 30 minutes through 3000 Hz- amplitude modulated frequency at once
Arm/Group | Zeltiq on Left | Electrical Stimulation on Right Side Thigh
Number analyzed (Participants) | 14 | 14
inches | 0.043 (0.0362) | -0.15 (0.1558)
Statistical Analysis 1: Comparison: Zeltiq on Left; Test type: Other; p = 0.503, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.669, Standard Deviation 0.03

3. Secondary Outcome: Change of the Fat Amount of Both Thighs Between Baseline and 12 Weeks
Description: The mean differences of the Cross-Sectional Areas of both Thighs between Baseline and 12 weeks
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- The Change of Fat on Left Thigh Between Baseline and 12 Weeks: Comparison of Cross-Sectional Area on Left Thigh by CT between baseline and 12 weeks
- The Change of Fat Right Thigh Between Baseline and 12 Weeks: Comparison of Cross-Sectional areas on Right thigh by CT between baseline and 12 weeks
Arm/Group | The Change of Fat on Left Thigh Between Baseline and 12 Weeks | The Change of Fat Right Thigh Between Baseline and 12 Weeks
Number analyzed (Participants) | 14 | 14
mm^2 | 1597.8853 (155.7977453) | 1970.0147 (398.15115)

4. Secondary Outcome: Change of Girths in Both Thighs for 12 Weeks
Description: Comparison of circumferences of both thighs for 12 weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: inch
Arm/Group | Zeltiq | Electrical Stimulation
Number analyzed (Participants) | 14 | 14
inch | -0.45 (0.17) | -0.15 (0.29)

5. Secondary Outcome: Weight Change for 12 Weeks
Description: Change in weight for 12 weeks
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Zeltiq | Electrical Stimulation
Number analyzed (Participants) | 14 | 14
Kg | -0.38 (0.81) | -0.38 (0.81)

ADVERSE EVENTS:
Groups:
- Electrical Stimulation: The radio frequency method was applied on right thigh (control side) as sham procedure for 30 minutes through 3000 Hz- amplitude modulated frequency at once.
Arm/Group | Zeltiq | Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 4/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zeltiq (N=14) | Electrical Stimulation (N=14)
Minor dermatological compliaint (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — pain
Minor Dermatologic complaint (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — bruits
Minor generalized complaints (Gastrointestinal disorders) | 1 (1) | 0 (0) — blood tinged stool

LIMITATIONS AND CAVEATS:
In the beginning, because this study has some drawback for small sample size , and secondly, although the novel treatment process for radio frequency method included more than 6 sessions, it was performed just at once as sham procedure in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No